CLINICAL TRIAL: NCT01630798
Title: A Phase 1B In-Vivo Esophageal Protocol for Detection of Neoplasia in the Digestive Tract
Brief Title: A In-Vivo Esophageal Protocol for Detection of Neoplasia in the Digestive Tract
Acronym: NTR 1B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Missy Tuck, Project Manager, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00062875
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Barrett's Esophagus
Keywords: barrett's esophgus; High grade dysplasia; Esophageal adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Application of peptide (Experimental)
  Interventions: Drug: GI heptapeptide

INTERVENTIONS:
Drug: GI heptapeptide — Investigational Agent Name: GI heptapeptide, Linear, 7 amino acid peptide sequence ASYNYDA with a 5-FITC tag and NH2 terminus. Investigational Agent Administration (see SOP in Appendix C) ASYNYDA-GGGSK-(5-FITC)-NH2 0.8 mg lyophilized powder per single-use amber vial Lyophilized powder reconstituted with 5 ml of 0.9% NaCl Final 100 µM concentration for single, one-time topical application Entire 5 ml volume (100 uM concentration) will be sprayed topically onto esophagus by the nurse/physician during the procedure through a standard endoscopy spray catheter (Olympus Medical, Tokyo Japan, PW-5V-1)

SUMMARY:
You are invited to participate in a research study to develop new ways to look for abnormal areas/tissues of the esophagus. The current endoscopes used to look at the esophagus are very good, but if the area doesn't look different to the naked eye, then the endoscope can't improve on that. The investigators are looking at using special fluorescent stains in addition to special endoscopes designed to see abnormal areas that are not obvious to the naked eye. Currently specialized microscopes and fluorescent stains are used in clinical laboratories but it takes several days of processing to get results. It may be very helpful to look for areas to sample for abnormal tissue during the endoscopy procedure.

You are being asked to let us use "fluorescent peptides" with a special endoscope that allow us to "see" your esophagus with both fluorescent and white light during your upper GI endoscopy procedure to help target your biopsies. Peptides are small chains of amino acids (the building blocks that make up proteins) linked together. Our peptide is a chain of 7 amino acids attached to a fluorescent dye called FITC (like the one used by your eye doctor).

The investigators have prepared special "fluorescent peptides", that will "glow" when a special light is used that should help us separate normal tissue from abnormal tissue. In this study, the investigators will apply the special fluorescent peptides by a spray catheter to your esophagus to help us target you biopsies. Both routine and targeted biopsies will be taken as your endoscopist feels is indicated.

This is a phase 1b study. This means that although the investigators have applied the peptide to 25 people in our first research study, the investigators still need to learn more about "fluorescent peptide" in people. The Food and Drug Administration (FDA) has not approved this agent, but is allowing us to test it in this study. The main goal of this study is to see if the peptide "glows" well and if the investigators can take pictures of the areas that do glow.

This is a research study of the peptide and our ability to see it "light up or fluoresce". Being in this study and applying this peptide won't change how your biopsies are taken nor how your endoscopy is done.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Barrett's Esophagus or esophageal adenocarcinoma with or without confirmed Barrett's Esophagus
* Subjects who are scheduled for a clinically-indicated upper endoscopic evaluation and/or intervention (e.g. esophagogastroduodenoscopy (EGD) with biopsies)
* All subjects who are medically cleared for the procedure (e.g. washout for anticoagulants, co-morbidities) who meet the inclusion/exclusion will be included. Standard practice guidelines for safely proceeding with the procedure will be sufficient for our study
* Adults aged 18 years to 100
* Willing and able to sign informed consent

Exclusion Criteria:

* Subjects with known allergy or negative reaction to fluorescein or derivatives
* Subjects who have had an esophagectomy
* Subjects who are also prepped for colonoscopy with the EGD
* Subjects on active chemotherapy or radiation treatment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
validate binding of the fluorescent-labeled peptide to esophageal neopla | 1.5 years
  The overall aim of this research project is to develop the use of fluorescent-labeled peptides that affinity bind to pre-cancerous mucosa in the digestive tract for use as an imaging agent to guide endoscopic biopsy or endoscopic mucosal resection (EMR). This particular study is a phase Ib, vaidation of efficacy of the topically applied peptide and continuing assessment of safety.
  To validate binding of the fluorescent-labeled peptide to esophageal neoplasia using an Olympus FITC Endoscopic Molecular Imaging System.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Kim Turgeon, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Joshi BP, Duan X, Kwon RS, Piraka C, Elmunzer BJ, Lu S, Rabinsky EF, Beer DG, Appelman HD, Owens SR, Kuick R, Doguchi N, Turgeon DK, Wang TD. Multimodal endoscope can quantify wide-field fluorescence detection of Barrett's neoplasia. Endoscopy. 2016 Feb;48(2):A1-A13. doi: 10.1055/s-0034-1392803. Epub 2015 Oct 1. PMID 26426999